CLINICAL TRIAL: NCT03472287
Title: A Multi-Center Study to Evaluate the Pharmacokinetics of Diacerein and Rhein and the Safety of Diacerein After Maximum Use, Topical Administration of CCP-020 (Diacerein 1% Ointment) to Patients With Epidermolysis Bullosa (EB)
Brief Title: To Evaluate the Pharmacokinetic of Diacerein and Rhein After Maximum Use in Patients With Epidermolysis Bullosa (EB)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Castle Creek Pharmaceuticals, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CCP-020-101
Record Dates: First submitted 2018-03-14; First posted 2018-03-21 (Actual); Results first posted 2020-02-10 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2020-02

CONDITIONS: Epidermolysis Bullosa (EB); Epidermolysis Bullosa Simplex; Dystrophic Epidermolysis Bullosa; Junctional Epidermolysis Bullosa
Keywords: EB; EBS; DEB; JEB
MeSH Terms: conditions — Epidermolysis Bullosa; Epidermolysis Bullosa Simplex; Epidermolysis Bullosa Dystrophica; Epidermolysis Bullosa, Junctional | interventions — diacerein; Ointments

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Adolescents, Adults) (Experimental): Adolescent and adult subjects with EB (aged 12 years and older) received diacerein 1% ointment daily for 10 days.
  Interventions: Drug: Diacerein 1% Ointment
- Cohort 2 (Children) (Experimental): Children with EB (aged 4 to 11 years, inclusive) received diacerein 1% ointment daily for 10 days.
  Interventions: Drug: Diacerein 1% Ointment

INTERVENTIONS:
Drug: Diacerein 1% Ointment — Diacerein 1% Ointment administered topically
  Other Names: CCP-020

SUMMARY:
A pharmacokinetic (PK) study in 16-20 EB subjects to be allocated to two cohorts. Cohort 1 to include 8-10 subjects (ages 12 yrs and older); Cohort 2 to include 8-10 subjects (ages 6 months-11 yrs, inclusive). Cohort 2 only included subjects 4 yrs and older. Serial PK blood sampling collected on Days 1 and 10. Analyses were performed to determine the concentrations of diacerein and rhein.

DETAILED DESCRIPTION:
This was an open-label, single-period study that intended to include subjects with EB consisting of infants/ children (ages 6 months to 11 years, inclusive) and adolescents/ adults (ages 12 years and older). The study included 2 cohorts.

Cohort 1 was to include adolescent/adult subjects with EB (ages 12 years and older);

Cohort 2 was to include infants/children with EB (ages 4 to 11 years, inclusive).

For both cohorts, the study intended to enroll subjects with epidermolysis bullosa simplex (EBS), dystrophic epidermolysis bullosa (DEB), and junctional epidermolysis bullosa (JEB) with lesions encompassing >/=2% BSA. The diacerein application area was >/=5% BSA and included lesioned and non-lesioned skin (if lesions accounted for <5% BSA); however, topical administration was </=30% BSA. On Days 1 and 10, the topical dose of study drug was applied by study staff, and blood was sampled for PK analyses of diacerein and rhein pre-dose and through 8 hours post-application. On Days 2 to 9, study drug was applied to the application area(s) at home. For Cohort 1, trough PK samples were collected on any 2 available days from Days 3 through 9, and study drug was applied after blood draw, while for Cohort 2 trough PK analyses were not performed.

ELIGIBILITY:
Key Inclusion Criteria:

* At least 12 years of age (Cohort 1) or at least 6 months of age to 11 years, inclusive (Cohort 2) at screening. For US only: at least 4 years of age to 11 years, inclusive (Cohort 2)
* The subject must weigh at least 9 kg (19.8 lbs) at Screening.
* Subject has a documented genetic mutation consistent with EB.
* Subject has EB lesions on ≥ 2% body surface area (BSA) and the EB lesions are in the following body areas: a. Localized: plantar and/or palmar areas, b. Generalized: arms, legs, torso, hands and feet.

Key Exclusion Criteria:

* Subject has EB lesions where drug will be applied that are infected
* Subject has used any diacerein containing product within 1 month prior to Visit 1
* Subject has used systemic immunotherapy or cytotoxic chemotherapy within 60 days prior to dosing.
* Subject has used systemic steroidal therapy or has used topical steroidal therapy on the EB lesions in the application area within 14 days prior to dosing
* Subject has participated in an investigational drug trial in which administration of an investigational study medication occurred within 30 days prior to dosing

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-05-18 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Spellman, Study Chair — Castle Creek Pharmaceuticals, LLC
Locations (3):
- United States (3):
  - Stanford School of Medicine, Palo Alto, California
  - Northwestern University Medical Center, Chicago, Illinois
  - UNC Dermatology, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1 (Adolescents, Adults): Adolescent and adult subjects with EB (aged 12 and older) received diacerein 1% ointment daily for 10 days
Period: Overall Study
Arm/Group | Cohort 1 (Adolescents, Adults) | Cohort 2 (Children)
Started | 8 | 3
Completed | 8 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1 (Adolescents, Adults): Adolescent and adult patients with EB (aged 12 and older) received Diacerein 1% Ointment daily for 10 days.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 (Adolescents, Adults) | Cohort 2 (Children) | Total
Number analyzed (Participants) | 8 | 3 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.5 (11.74) | 8.3 (1.53) | 21.5 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 6
  Male | 3 | 2 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 7 | 1 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 7 | 2 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 3 | 11
EB Classification per Cohort [Number; unit: participants]
  Epidermolysis Bullosa Simplex (EBS) | 4 | 3 | 7
  Dystrophic Epidermolysis Bullosa (DEB) | 4 | 0 | 4
  Junctional Epidermolysis Bullosa (JEB) | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Detectable Plasma Concentrations of Diacerein and Rhein
Description: Bioanalytical analyses were performed to determine concentrations levels of diacerein and rhein in plasma using validated bioanalytical methods.
  For Cohort 1, blood samples were taken at pre-dose and 0.5, 1, 2, 3, 4, 6, and 8 hours post-dose.
  For Cohort 2, blood samples were taken at pre-dose and 1, 2, 4, 6, and 8 hours post-dose.
  Trough PK samples were collected on any 2 available days from Days 3 through 9 for Cohort 1 only.
  Summary statistics for each scheduled time were only reported if at least 50% of subjects had quantifiable concentrations.
Time Frame: Days 1-10, at select time points per protocol
Population: Cohort 1: 4 adolescent/adult subjects with EBS, 4 adolescent/adult subjects with DEB; Cohort 2: 3 child subjects with EBS
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1 (Adolescents, Adults): Adolescent/adult subjects with EB (aged 12 years and older) received diacerein 1% ointment daily for 10 days.
- Cohort 2 (Children): Children with EB (ages 4-11 yrs, inclusive) were administered diacerein 1% ointment topically for 10 days.
Arm/Group | Cohort 1 (Adolescents, Adults) | Cohort 2 (Children)
Number analyzed (Participants) | 8 | 3
Participants
  Rhein Below the limit of quantification:EBS: number analyzed (Participants) | 4 | 3
  Rhein Below the limit of quantification:EBS | 3 | 2
  Rhein Below the limit of quantification:DEB: number analyzed (Participants) | 4 | 0
  Rhein Below the limit of quantification:DEB | 0 | 0
  Rhein Above Lower limit of quantification:EBS: number analyzed (Participants) | 4 | 3
  Rhein Above Lower limit of quantification:EBS | 1 | 1
  Rhein Above Lower limit of quantification:DEB: number analyzed (Participants) | 4 | 0
  Rhein Above Lower limit of quantification:DEB | 4 | 0
  Diacerein Below the limit of quantification:EBS: number analyzed (Participants) | 4 | 3
  Diacerein Below the limit of quantification:EBS | 4 | 3
  Diacerein Below the limit of quantification:DEB: number analyzed (Participants) | 4 | 0
  Diacerein Below the limit of quantification:DEB | 4 | 0
  Diacerein Above Lower limit of quantification:EBS: number analyzed (Participants) | 4 | 3
  Diacerein Above Lower limit of quantification:EBS | 0 | 0
  Diacerein Above Lower limit of quantification:DEB: number analyzed (Participants) | 4 | 0
  Diacerein Above Lower limit of quantification:DEB | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline to 30 days after last dose of study drug application (40 days)
Groups:
- Cohort 1 (Adolescents, Adults): Adolescent/adult patients with EB (aged 12 and older) received Diacerein 1% Ointment daily for 10 days
Arm/Group | Cohort 1 (Adolescents, Adults) | Cohort 2 (Children)
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/3
Other Adverse Events (participants affected / at risk) | 1/8 | 0/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (Adolescents, Adults) (N=8) | Cohort 2 (Children) (N=3)
Pyrexia (General disorders) | 1 (1) | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-01-07): https://cdn.clinicaltrials.gov/large-docs/87/NCT03472287/SAP_000.pdf
  • Study Protocol (2018-02-07): https://cdn.clinicaltrials.gov/large-docs/87/NCT03472287/Prot_001.pdf